CLINICAL TRIAL: NCT07151404
Title: Efficacy of Acupuncture at Lieque (LU7) Based on Six Command Points Theory, Combined With Electroacupuncture at Jiaji (Ex-B2, C4-C7) and Cervical-Shoulder Points in Cervical Spondylosis
Brief Title: Efficacy of Acupuncture at Lieque (LU7) for Neck Pain in Cervical Spondylosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nguyen Ngoc Doan Thuy (Other)
Responsible Party: Sponsor-Investigator, Nguyen Ngoc Doan Thuy, MSc, MD, Lecturer, Department of Acupuncture, School of Medicine - Vietnam National University at Ho Chi Minh City, School of Medicine - Vietnam National University at Ho Chi Minh city
Organization: School of Medicine - Vietnam National University at Ho Chi Minh city (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C2025-44-13; 86/QĐ-ĐHQG (Other Grant/Funding Number: Vietnam National University, Ho Chi Minh City)
Record Dates: First submitted 2025-08-19; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cervical Spondylosis; Neck Pain
Keywords: Cervical Spondylosis; Neck Pain; Cervical Spine; Acupuncture; Electroacupuncture; Lieque Point; LU7 Acupoint; Jiaji Points; Cervical-Shoulder Acupoints; Randomized Controlled Trial; LU7; Ex-B2; Ex-B2, C4-C7
MeSH Terms: conditions — Spondylosis; Neck Pain | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two groups. The experimental group will receive filiform needle acupuncture at Lieque (LU7) combined with electroacupuncture at Jiaji (Ex-B2, C4-C7) and selected neck-shoulder acupoints. The control group will receive electroacupuncture at Jiaji (Ex-B2, C4-C7) and neck-shoulder acupoints only. Treatment will be performed once daily for a total of 20 sessions over approximately 4 weeks, excluding Sundays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lieque (LU7) + Electroacupuncture (Experimental): Participants will receive filiform needle acupuncture at Lieque (LU7) combined with electroacupuncture at Jiaji (Ex-B2, C4-C7) and neck-shoulder acupoints. Sterile disposable filiform needles (0.3 × 25 mm) will be used. Electroacupuncture will be applied at 60 Hz continuous wave for 30 minutes per session. Treatment will be given once daily for a total of 20 sessions, excluding Sundays (approximately 4 weeks).
  Interventions: Procedure: Acupuncture at LU7 (Lieque) + Electroacupuncture
- Electroacupuncture Only (Active Comparator): Participants will receive electroacupuncture at Jiaji (Ex-B2, C4-C7) and neck-shoulder acupoints only, without acupuncture at Lieque (LU7). Electroacupuncture will be applied at 60 Hz continuous wave for 30 minutes per session. Treatment will be given once daily for a total of 20 sessions, excluding Sundays (approximately 4 weeks).
  Interventions: Procedure: Electroacupuncture Only

INTERVENTIONS:
Procedure: Acupuncture at LU7 (Lieque) + Electroacupuncture — Participants will receive filiform needle acupuncture at Lieque (LU7) combined with electroacupuncture at Jiaji (Ex-B2, C4-C7) and neck-shoulder acupoints including Fengchi (GB20), Jianjing (GB21), Tianzhu (BL10), and Dazhu (BL11). Sterile disposable filiform needles (0.3 × 25 mm) will be inserted at LU7 using standard manual acupuncture technique. Electroacupuncture will be delivered with continuous wave stimulation at 60 Hz for 30 minutes per session. Treatment will be performed once daily for a total of 20 sessions over approximately 4 weeks, excluding Sundays.
  Other Names: Filiform Needle Acupuncture at Lieque (LU7); Filiform Needle Acupuncture at LU7; Filiform Needle Acupuncture
  Arms: Lieque (LU7) + Electroacupuncture
Procedure: Electroacupuncture Only — Participants will receive electroacupuncture at Jiaji (Ex-B2, C4-C7) and neck-shoulder acupoints including Fengchi (GB20), Jianjing (GB21), Tianzhu (BL10), and Dazhu (BL11), without acupuncture at Lieque (LU7). Electroacupuncture will be delivered with continuous wave stimulation at 60 Hz for 30 minutes per session. Treatment will be performed once daily for a total of 20 sessions over approximately 4 weeks, excluding Sundays.
  Other Names: Electroacupuncture; Electroacupuncture Control; EA at Jiaji and Neck-Shoulder Acupoints; EA; Electroacupuncture at Jiaji and Neck-Shoulder Acupoints
  Arms: Electroacupuncture Only

SUMMARY:
Cervical spondylosis is a common degenerative disorder of the cervical spine that often leads to chronic neck pain, stiffness, and reduced daily functioning. Pain management in these patients remains challenging, and acupuncture is widely used as a non-pharmacological treatment option. However, the additional benefit of stimulating the Lieque (LU7) acupoint, based on the Six Command Points theory, has not been fully established.

This randomized controlled trial will evaluate whether acupuncture at Lieque (LU7), combined with electroacupuncture at Jiaji (Ex-B2, C4-C7) and cervical-shoulder points, provides greater pain relief compared to electroacupuncture at Jiaji (Ex-B2, C4-C7) and cervical-shoulder points alone.

A total of 130 participants with cervical spondylosis will be randomly assigned to two groups. Treatments will be delivered over 20 days. The primary outcome is the change in neck pain intensity, measured by a 0-100 mm Visual Analog Scale (VAS), from baseline to the end of treatment.

The findings will provide clinical evidence on the effectiveness of acupuncture at Lieque (LU7) for reducing neck pain and improving patient outcomes in cervical spondylosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Diagnosis of cervical spondylosis based on clinical evaluation and imaging.
* Presence of cervical spine syndrome, including:

  * Neck and shoulder pain.
  * Limited range of motion in the cervical spine.
  * Local tenderness over the cervical spine or paraspinal region corresponding to nerve roots.
* Radiographic evidence of cervical spondylosis on standard X-ray (frontal, lateral, or oblique views), showing one or more of the following:

  * Subchondral sclerosis.
  * Narrowing of the intervertebral disc space.
  * Osteophyte formation (bone spurs, bridging osteophytes).
* Patients receiving treatment at Thu Duc City Hospital

Exclusion Criteria:

* Patients who do not agree to participate in the study.
* Acute torticollis, cervical disc herniation, spinal deformity, cervical spine trauma, or spinal tumors.
* Neck and shoulder pain not caused by cervical spondylosis.
* History of systemic diseases such as rheumatoid arthritis, severe cardiovascular disease, systemic infection, malignancy, or immunodeficiency disorders.
* History of neurological or psychiatric conditions that impair communication or compliance, including speech disorders, impaired consciousness, psychosis, or dementia.
* Contraindications to electroacupuncture.
* Non-compliance with study treatment protocol.
* Use of non-steroidal anti-inflammatory drugs (NSAIDs) within the past 10 days or local corticosteroid injection within the past 3 months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Neck Pain Intensity (VAS Score) | Baseline (D0), Day 10 (D10), and Day 20 (D20).
  Pain intensity in the neck region will be assessed using a 100-mm Visual Analogue Scale (VAS), where 0 mm = no pain and 100 mm = worst possible pain.

SECONDARY OUTCOMES:
Change in Neck Pain Questionnaire (NPQ) Score | Baseline (D0), Day 10 (D10), and Day 20 (D20).
  The NPQ (8-item version) will be used to assess disability related to neck pain. It covers 8 domains: pain intensity, pain and sleep, nocturnal paresthesia, duration of symptoms, carrying objects, reading/TV, work/housework, and social activities. Each domain is scored 0-4; total score ranges from 0 (no disability) to 32 (severe disability). Higher scores indicate greater disability.
Change in Cervical Range of Motion (ROM) | Baseline (D0), Day 10 (D10), and Day 20 (D20).
  Cervical spine ROM (flexion, extension, right/left lateral flexion, right/left rotation) will be measured in degrees using a goniometer (or inclinometer). Higher values indicate greater mobility.

OTHER OUTCOMES:
Adverse Events Related to Acupuncture/Electroacupuncture | Throughout the 20 treatment sessions (approximately 4 weeks).
  All adverse events will be systematically recorded, including but not limited to: nausea, fatigue, dizziness, heavy numbness of the limbs, and other unexpected events. Each event will be assessed for severity (mild, moderate, severe) and its possible relationship to the intervention.
Distribution of Traditional Chinese Medicine (TCM) Syndrome Types | At baseline (D0), prior to intervention.
  Participants will be classified into Traditional Chinese Medicine (TCM) syndromes according to TCM diagnostic criteria:
  Wind-Cold-Damp Bi Syndrome (WCDBS) Wind-Damp-Heat Bi Syndrome (WDHBS) Qi Stagnation and Blood Stasis (QSBS) Liver and Kidney Yin Deficiency (LKYD) The frequency and proportion of each syndrome type will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ngoc Doan Thuy Nguyen, MD, MSc, Principal Investigator — University of Health Sciences, Vietnam National University Ho Chi Minh City
Locations (1):
- Thu Duc City Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to concerns regarding data confidentiality and patient privacy.